CLINICAL TRIAL: NCT02836093
Title: Pilot Study for Assessment of Exercise Capacity in Breast Cancer Patients With Radiotherapy-Related Fatigue
Brief Title: Exercise Testing for Early Stage Breast Cancer Patients Receiving Radiation Treatment
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-941
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer; Fatigue
Keywords: Exercise; Radiation Treatment; 16-941
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- evaluations/assessments
  Interventions: Behavioral: FACIT-Fatigue 52-point questionnaire

INTERVENTIONS:
Behavioral: FACIT-Fatigue 52-point questionnaire

SUMMARY:
Many patients receiving radiation therapy for breast cancer experience fatigue although doctors do not fully understand why. The purpose of this study is to test if patients who experience fatigue during radiation treatment for breast cancer have changes in their capability to perform exercise on a treadmill.

ELIGIBILITY:
Inclusion Criteria:

* Female
* ECOG performance status 0 or 1
* Medical clearance from attending radiation oncologist or medical oncologist to undergo a symptom-limited CPET
* Currently undergoing intact breast radiotherapy for early stage breast cancer (including TisN0, T1N0, T2N0) or has completed intact breast RT in the last 3 months.
* Receiving or received a prescribed dose of 4240 cGy in 16 fractions to the whole breast without treatment directed at nodal basins. Patients may also be receiving or have received a boost to the lumpectomy bed at the discretion of the treating physician.
* Subjects may be treated in the supine or prone position at the discretion of the treating physician.
* Subjects may be treated with or without a deep inspiratory breath hold technique at the discretion of the treating physician.
* Identified by the treating radiation oncologist as having significant treatment-related fatigue or minimal treatment-related fatigue and not simply baseline fatigue. A score of "0" on the RTOG fatigue scale will be considered minimal fatigue, while a score of "2" or greater will be considered significant fatigue (moderate fatigue causing difficulty performing some ADLs).

Exclusion Criteria:

* Currently undergoing post-mastectomy radiation
* Has received chemotherapy previously or has a plan to receive chemotherapy during the timeframe of study assessment.
* Any of the following absolute contraindications to CPET, as per American Thoracic Society (ATS) recommendations

  * Acute myocardial infarction (within 3-5 days of any planned study procedures)
  * Unstable angina
  * Uncontrolled arrhythmia causing symptoms or hemodynamic compromise
  * Recurrent syncope
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Symptomatic severe aortic stenosis
  * Uncontrolled heart failure
  * Acute pulmonary embolus or pulmonary infarction within 3 months of any planned study procedures
  * Thrombosis of lower extremities
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Pulmonary edema
  * Room air desaturation at rest ≤ 85%
  * Respiratory failure
  * Acute non-cardiopulmonary disorders that may affect exercise performance or be aggravated by exercise (i.e. infection, renal failure, thyrotoxicosis)
  * Mental impairment leading to inability to cooperate

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing or have recently completed radiotherapy for breast cancer (in the last 3 months) will be assessed in outpatient clinics of the Radiation Oncology Department of MSKCC. The protocol is available for consenting only at OneMSK Sites Basking Ridge, Rockville Center, Commack, Monmouth and Westchester.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
fatigue measurement using the 13-item FACIT-fatigue scale | 1 year
  Fatigue will be assessed using the 13-item FACIT-fatigue scale for the assessment of fatigue in cancer patients.24 The FACIT-Fatigue is a validated questionnaire that was originally developed for the precise evaluation of fatigue levels in cancer patients with anemia. It consists of 13 questions using a 5 point scale (0=not at all; 1 = a little bit, 2 = somewhat, 3 = quite a bit and 4 = very much). It has been used frequently in the clinical trial setting (please see appendix 1). Responses to each question are added with equal weight to obtain a total score. The range of possible scores is 0-52, with 0 corresponding to the highest level of fatigue and 52 corresponding to the lowest level of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Beryl McCormick, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre (Consent only), Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/